CLINICAL TRIAL: NCT02607306
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide, Insulin Degludec and Liraglutide in Japanese Subjects With Type 2 Diabetes Mellitus
Acronym: DUAL™ I Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-4183; U1111-1170-1332 (Other: WHO); JapicCTI-153089 (Other: JAPIC)
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Results first posted 2019-07-29 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Insulin degludec/liraglutide OD (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Insulin degludec OD (Active Comparator)
  Interventions: Drug: insulin degludec
- Liraglutide OD (Active Comparator)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Injected s.c. / subcutaneously (under the skin) once daily (OD) , in combination with pre-trial OAD (oral antidiabetic drug)kept in unchanged dose.
  Arms: Insulin degludec/liraglutide OD
Drug: insulin degludec — Injected s.c. / subcutaneously (under the skin) once daily (OD) , in combination with pre-trial OAD (oral antidiabetic drug)kept in unchanged dose.
  Arms: Insulin degludec OD
Drug: liraglutide — Injected s.c. / subcutaneously (under the skin) once daily (OD) , in combination with pre-trial OAD (oral antidiabetic drug)kept in unchanged dose.
  Arms: Liraglutide OD

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare the efficacy and safety of insulin degludec/liraglutide, insulin degludec and liraglutide in Japanese subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese subjects, age at least 20 years at the time of signing informed consent
* Type 2 diabetes subjects (diagnosed clinically) at least 6 months prior to screening
* HbA1c (glycosylated haemoglobin) 7.0-11.0 % (both inclusive) by central laboratory analysis, with the aim of a median of 8.3%. When approximately 50% of the randomised subjects have a HbA1c above 8.3%, the remaining subjects randomised must have a HbA1c below or equal to 8.3%; or when approximately 50% of the randomised subjects have a HbA1c below or equal to 8.3%, the remaining subjects randomised must have a HbA1c above 8.3%
* Body-mass index (BMI) above or equal to 20 kg/m^2
* Subjects on stable therapy with one OAD (defined as unchanged medication and unchanged dose) for at least 60 days (metformin, a-GI, TZD, SU, SGLT2i or glinide) prior to screening according to approved Japanese labelling

Exclusion Criteria:

* Previous treatment with insulin (except for short-term treatment in connection with intercurrent illness including gestational diabetes)
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 60 days before screening
* Anticipated initiation or change in concomitant medications in excess of 14 days known to affect weight or glucose metabolism
* Impaired liver function, defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) equal to or above 2.5 times upper limit of normal
* Renal impairment estimated Glomerular Filtration Rate (eGFR) below 60mL/min/1.73m^2 as per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* Screening calcitonin equal to or above 50 ng/L
* History of pancreatitis (acute or chronic)
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN 2)
* Subjects presently classified as being in New York Heart Association (NYHA) Class IV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- Japan (63):
  - Novo Nordisk Investigational Site, Adachi-ku, Tokyo
  - Novo Nordisk Investigational Site, Akita-shi, Akita
  - Novo Nordisk Investigational Site, Annaka-shi, Gunma
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Chiba-shi, Chiba
  - Novo Nordisk Investigational Site, Chitose, Hokkaido
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Chuo-ku,Tokyo
  - Novo Nordisk Investigational Site, Chūōku
  - Novo Nordisk Investigational Site, Edogawa-ku, Tokyo
  - Novo Nordisk Investigational Site, Fujisawa-shi, Kanagawa
  - Novo Nordisk Investigational Site, Fukuoka-shi, Fukuoka
  - Novo Nordisk Investigational Site, Fukushima
  - Novo Nordisk Investigational Site, Gunma
  - Novo Nordisk Investigational Site, Hachioji-shi, Tokyo
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Ichihara-shi, Chiba
  - Novo Nordisk Investigational Site, Iruma-shi, Saitama
  - Novo Nordisk Investigational Site, Itabashi-ku, Tokyo
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Izumisano-shi,Osaka
  - Novo Nordisk Investigational Site, Kagoshima-shi, Kagoshima
  - Novo Nordisk Investigational Site, Kamakura-shi
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kanra-gun, Gunma
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Kawaguchi-shi, Saitama
  - Novo Nordisk Investigational Site, Kawasaki-shi,Kanagawa
  - Novo Nordisk Investigational Site, Kisarazu-shi, Chiba
  - Novo Nordisk Investigational Site, Kobe-shi, Hyogo
  - Novo Nordisk Investigational Site, Kuki-shi, Saitama
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Kushiro-shi, Hokkaido
  - Novo Nordisk Investigational Site, Kyoto-shi, Kyoto
  - Novo Nordisk Investigational Site, Minato-ku, Tokyo
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miura-shi, Kanagawa
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Obihiro-shi, Hokkaido
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Onga-gun, Fukuoka
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Saijo-shi, Ehime
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shizuoka-shi, Shizuoka
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Toshima-ku, Tokyo
  - Novo Nordisk Investigational Site, Toyonaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ube-shi, Yamaguchi
  - Novo Nordisk Investigational Site, Urasoe-shi,
  - Novo Nordisk Investigational Site, Yamaguchi-shi, Yamaguchi
  - Novo Nordisk Investigational Site, Yamato-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Kaku K, Araki E, Tanizawa Y, Ross Agner B, Nishida T, Ranthe M, Inagaki N. Superior efficacy with a fixed-ratio combination of insulin degludec and liraglutide (IDegLira) compared with insulin degludec and liraglutide in insulin-naive Japanese patients with type 2 diabetes in a phase 3, open-label, randomized trial. Diabetes Obes Metab. 2019 Dec;21(12):2674-2683. doi: 10.1111/dom.13856. Epub 2019 Aug 28. PMID 31407845
- [Result] Komatsu M, Watada H, Kaneko S, Ross Agner BF, Nishida T, Kaku K. Efficacy and safety of the fixed-ratio combination of insulin degludec and liraglutide by baseline glycated hemoglobin, body mass index and age in Japanese individuals with type 2 diabetes: A subgroup analysis of two phase III trials. J Diabetes Investig. 2021 Sep;12(9):1610-1618. doi: 10.1111/jdi.13525. Epub 2021 Mar 24. PMID 33595901
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 71 sites in Japan. 71 sites screened and randomised subjects.
Groups:
- Insulin Degludec/Liraglutide: Eligible subjects were treated with insulin degludec/liraglutide (IDegLira) once daily (OD) in combination with pre-trial oral anti diabetic drugs (at stable dose level and dosing frequency; dose reduction was allowed in case of safety concern). The recommended starting dose of IDegLira was 10 dose steps (10 units IDeg/0.36 mg liraglutide). IDegLira was titrated twice weekly according to a predefined titration algorithm to a maximum of 50 dose steps (50 units IDeg/1.8 mg liraglutide), aiming to reach a fasting plasma glucose target between 72 mg/dL (4.0 mmol/L) and 90 mg/dL (5.0 mmol/L). One follow-up visit was scheduled 7 days after end of treatment. IDegLira was injected subcutaneously in the thigh, upper arm (deltoid region) or abdomen. The injection area chosen remained unchanged throughout the trial, although rotation within the area was recommended.
- Insulin Degludec: Eligible subjects were treated with insulin degludec (IDeg) once daily (OD) in combination with pre-trial oral anti diabetic drugs (at stable dose level and dosing frequency unless there were safety concerns, in which case dose reduction was allowed). The recommended starting dose of IDeg was 10 units. IDeg was titrated twice weekly according to a predefined titration algorithm, aiming to reach a fasting plasma glucose target between 72 mg/dL (4.0 mmol/L) and 90 mg/dL (5.0 mmol/L). There was no maximum dose decided for IDeg. One follow-up visit was scheduled 7 days after end of treatment. IDeg was injected subcutaneously in the thigh, upper arm (deltoid region) or abdomen. The injection area chosen remained unchanged throughout the trial, although rotation within the area was recommended.
- Liraglutide: Eligible subjects were treated with liraglutide once daily (OD) in combination with pre-trial oral anti diabetic drugs (at stable dose level and dosing frequency unless there were safety concerns, in which case dose reduction was allowed). For liraglutide the starting dose of liraglutide was 0.3 mg/day and subsequent weekly dose escalation by 0.3 mg weekly to a fixed maximum dose of 1.8 mg/day. One follow-up visit was scheduled 7 days after end of treatment. Liraglutide was injected subcutaneously in the thigh, upper arm (deltoid region) or abdomen. The injection area chosen remained unchanged throughout the trial, although rotation within the area was recommended.
Period: Overall Study
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Started | 275 | 271 | 273
Completed | 254 | 248 | 263
Not Completed | 21 | 23 | 10
Not completed — Adverse Event | 8 | 6 | 6
Not completed — Unclassified | 1 | 4 | 0
Not completed — Withdrawal by Subject | 8 | 10 | 2
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Protocol Violation | 4 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide | Total
Number analyzed (Participants) | 275 | 271 | 273 | 819
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (10.2) | 57.8 (9.9) | 56.8 (10.1) | 57.2 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 76 | 81 | 238
  Male | 194 | 195 | 192 | 581
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 275 | 271 | 273 | 819
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 275 | 271 | 273 | 819
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.52 (1.12) | 8.53 (1.05) | 8.32 (0.99) | 8.45 (1.06)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin) Tested for Non-inferiority of IDegLira vs IDeg and Superiority of IDegLira vs Lira
Description: Change from baseline (week 0) in HbA1c after 52 weeks of treatment was measured. Statistical analyses were performed to test the hypotheses: non-inferiority of IDegLira vs. IDeg and superiority of IDegLira vs. Liraglutide (Lira).
Time Frame: Week 0, Week 52
Population: Full Analysis Set (FAS) included all randomised subjects (819 subjects). The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Missing data were imputed using last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Percentage of HbA1c | -2.42 (1.04) | -1.80 (1.02) | -1.80 (0.92)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Degludec; The change from baseline in response after 52 weeks are analysed using an ANCOVA model with treatment and pre-trial OAD as fixed factors and baseline HbA1c value as covariate; Test type: Non-Inferiority — Non-inferiority of IDegLira vs. IDeg was confirmed if the 95% confidence interval for the mean treatment difference lies entirely below 0.3%; p < 0.0001, ANCOVA — p-value for non-inferiority of IDegLira vs IDeg is presented; Treatment contrast = -0.63, 95% CI 2-sided [-0.75 to -0.52]
Statistical Analysis 2: Comparison: Insulin Degludec/Liraglutide vs Liraglutide; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Superiority of IDegLira vs. Lira was confirmed if the 95% confidence interval for the mean treatment difference for change from baseline in HbA1c lies entirely below 0.0%; p < 0.0001, ANCOVA — p-value for superiority of IDegLira vs Lira is presented; Treatment contrast = -0.48, 95% CI 2-sided [-0.60 to -0.37]

2. Secondary Outcome: Change From Baseline in Body Weight (kg)
Description: Change from baseline (week 0) in body weight after 52 weeks of treatment.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Kg | 2.9 (3.2) | 4.1 (4.3) | -1.0 (3.4)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Degludec; The change from baseline in response after 52 weeks were analysed using an ANCOVA method with treatment and pre-trial OAD treatment as fixed factors and baseline body weight as covariate; Test type: Superiority — A hierarchical testing procedure is used to control the overall type I error on a two sided 5% level. If and only if non-inferiority of IDegLira vs. IDeg and superiority of IDegLira vs. Lira are confirmed in the primary analysis (change in HbA1c), the three secondary confirmatory tests are performed for superiority of IDegLira versus IDeg with a fixed sequence (1. change in body weight, 2. number of treatment emergent severe or BG confirmed hypoglycaemic episodes and 3. change in HbA1c); p = 0.0001, ANCOVA — p-value for superiority of IDegLira vs IDeg is presented; Treatment contrast = -1.19, 95% CI 2-sided [-1.80 to -0.59]

3. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose (BG) Confirmed Hypoglycaemic Episodes
Description: Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with or without symptoms consistent with hypoglycaemia.
  Severe hypoglycaemia according to the ADA definition: an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: Weeks 0-52
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (819 subjects). Subjects in the safety set contributed to the evaluation "as treated".
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Episodes | 467 | 869 | 13
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Degludec; The number of events is analysed using a negative binomial regression model (log link) with the logarithm of the treatment emergent exposure time (100 years) as offset. The model includes treatment and pre-trial OAD treatment as fixed factors; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Negative binomial regression — p-value for superiority of IDegLira vs IDeg is presented; Treatment contrast = 0.48, 95% CI 2-sided [0.35 to 0.68]

4. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin) Tested for Superiority of IDegLira vs IDeg
Description: Change from baseline (week 0) in HbA1c after 52 weeks of treatment was measured. Statistical analysis was performed to test the hypothesis: superiority of IDegLira vs. IDeg.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Percentage of HbA1c | -2.42 (1.04) | -1.80 (1.02) | -1.80 (0.92)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Degludec; The change from baseline in response after 52 weeks are analysed using an ANCOVA model with treatment, pre-trial OAD as fixed factors and corresponding baseline HbA1c value as covariate; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, ANCOVA — p-value for superiority of IDegLira vs IDeg is presented; Treatment contrast = -0.63, 95% CI 2-sided [-0.75 to -0.52]

5. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in FPG after 52 weeks
Time Frame: Week 0, Week 52
Population: Full Analysis Set (FAS) included all randomised subjects (819 subjects). The statistical evaluation of the FAS followed the intention-to-treat (ITT) principle and subjects contributed to the evaluation "as randomised". Missing data were imputed using last observation carried forward (LOCF) method. Number Analyzed = subjects with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 272
mmol/L | -4.08 (2.47) | -3.97 (2.56) | -2.62 (1.95)

6. Secondary Outcome: Insulin Dose
Description: Actual daily total insulin dose after 52 weeks of treatment.
Time Frame: After 52 weeks of treatment
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (819 subjects). Subjects in the safety set contributed to the evaluation "as treated". Missing data were imputed using LOCF method. This endpoint evaluation is only applicable for subjects in IDegLira and IDeg arm.
Measure: Mean (Standard Deviation); unit: Insulin Units/Day
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 275 | 271
Insulin Units/Day | 27.7 (14.8) | 34.8 (26.0)

7. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0%
Description: Number of subjects with HbA1c less than 7.0% after 52 weeks of treatment.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Participants
  Yes | 245 | 189 | 208
  No | 30 | 82 | 65

8. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0% and Change in Body Weight From Baseline Below or Equal to Zero
Description: Number of subjects with HbA1c less than 7.0% and without weight gain after 52 weeks of treatment.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Participants
  Yes | 44 | 22 | 142
  No | 231 | 249 | 131

9. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0% Without Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment.
Description: Number of subjects with HbA1c less than 7.0% after 52 weeks, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 52 weeks of treatment
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 270 | 265 | 271
Participants
  Yes | 227 | 169 | 206
  No | 43 | 96 | 65

10. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 7.0% and Change in Body Weight From Baseline Below or Equal to Zero and Without Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: Number of subjects with HbA1c less than 7.0% and without weight gain, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 52 weeks of treatment
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 270 | 265 | 271
Participants
  Yes | 37 | 22 | 141
  No | 233 | 243 | 130

11. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 6.5%
Description: Number of subjects with HbA1c less than 6.5% after 52 weeks of treatment.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Participants
  Yes | 213 | 134 | 171
  No | 62 | 137 | 102

12. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 6.5% and Change in Body Weight From Baseline Below or Equal to Zero
Description: Number of subjects with HbA1c less than 6.5% and without weight gain after 52 weeks of treatment.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Participants
  Yes | 41 | 17 | 126
  No | 234 | 254 | 147

13. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 6.5% Without Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment.
Description: Number of subjects with HbA1c less than 6.5% after 52 weeks, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 52 weeks of treatment
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 270 | 265 | 271
Participants
  Yes | 198 | 123 | 170
  No | 72 | 142 | 101

14. Secondary Outcome: Responder (Yes/no): HbA1c Less Than 6.5% and Change in Body Weight From Baseline Below or Equal to Zero and Without Treatment Emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes During the Last 12 Weeks of Treatment
Description: Number of subjects with HbA1c less than 6.5% with no weight gain, who did not experience treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes during the last 12 weeks of treatment.
  Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: After 52 weeks of treatment
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 270 | 265 | 271
Participants
  Yes | 35 | 17 | 125
  No | 235 | 248 | 146

15. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference after 52 weeks of treatment.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cm
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Cm | 2.5 (4.5) | 3.4 (5.2) | -1.1 (4.4)

16. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic)
Description: Change from baseline in blood pressure (systolic and diastolic) after 52 weeks of treatment.
Time Frame: Week 0, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
mmHg
  Systolic blood pressure | 1.7 (12.0) | 3.4 (14.3) | -1.8 (13.0)
  Diastolic blood pressure | 0.5 (7.9) | 0.6 (9.3) | -0.4 (8.3)

17. Secondary Outcome: Self-Measured Blood Glucose (SMBG) 9-point Profile: 9-point Profile (Individual Points in the Profile)
Description: Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime, at 4:00 a.m. and before breakfast the following day.
Time Frame: After 52 weeks of the treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
mmol/L
  Before breakfast | 5.90 (1.45) | 5.93 (1.64) | 7.35 (1.70)
  90 minutes after start of breakfast: number analyzed (Participants) | 274 | 271 | 272
  90 minutes after start of breakfast | 9.57 (2.83) | 10.43 (3.16) | 10.59 (3.25)
  Before lunch: number analyzed (Participants) | 275 | 269 | 270
  Before lunch | 6.01 (1.90) | 6.72 (2.59) | 6.87 (2.07)
  90 minutes after start of lunch: number analyzed (Participants) | 274 | 270 | 270
  90 minutes after start of lunch | 9.85 (3.16) | 11.12 (3.04) | 10.59 (3.38)
  Before dinner: number analyzed (Participants) | 274 | 271 | 273
  Before dinner | 6.47 (2.44) | 6.90 (2.57) | 7.03 (2.04)
  90 minutes after start of dinner: number analyzed (Participants) | 274 | 270 | 270
  90 minutes after start of dinner | 9.67 (3.01) | 10.89 (3.25) | 10.14 (3.03)
  Bedtime: number analyzed (Participants) | 271 | 269 | 268
  Bedtime | 8.27 (2.79) | 9.49 (3.28) | 8.73 (2.58)
  At 4:00 a.m.: number analyzed (Participants) | 272 | 268 | 270
  At 4:00 a.m. | 6.12 (1.70) | 6.41 (2.18) | 7.27 (1.79)
  Before breakfast the following day | 5.77 (1.56) | 5.71 (1.68) | 7.13 (1.68)

18. Secondary Outcome: Change in SMBG 9-point Profile - Mean of the 9-point Profile
Description: Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime, at 4:00 a.m. and before breakfast the following day. Mean of the 9-point profile was defined as the area under the profile (calculated using the trapezoidal method) divided by the measurement time.
Time Frame: Week 0, week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 269 | 272
mmol/L | -4.60 (2.65) | -3.84 (2.63) | -3.46 (2.37)

19. Secondary Outcome: Change in SMBG 9-point Profile - Mean of Postprandial Increments (From Before Meal to 90 Min After for Breakfast, Lunch and Dinner)
Description: Subjects were instructed to measure their plasma glucose at following timepoints: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, at bedtime, at 4:00 a.m. and before breakfast the following day. The mean increment over all meals was derived as the mean of all available meal increments.
Time Frame: Week 0, week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 269 | 272
mmol/L | -0.74 (2.51) | -0.27 (2.39) | -1.01 (2.38)

20. Secondary Outcome: Total Cholesterol as a Ratio to Baseline at 52 Weeks
Description: Total cholesterol after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Ratio | 0.92 (13.9) | 0.97 (11.9) | 0.94 (13.0)

21. Secondary Outcome: Low Density Lipoprotein (LDL) Cholesterol as a Ratio to Baseline at 52 Weeks
Description: Low density lipoprotein (LDL) cholesterol after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Ratio | 0.91 (23.4) | 0.99 (18.2) | 0.93 (24.2)

22. Secondary Outcome: High Density Lipoprotein (HDL) Cholesterol as a Ratio to Baseline at 52 Weeks
Description: High density lipoprotein (HDL) cholesterol after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Ratio | 0.94 (16.4) | 0.94 (14.6) | 0.99 (14.5)

23. Secondary Outcome: Very Low Density Lipoprotein (VLDL) Cholesterol as a Ratio to Baseline at 52 Weeks
Description: Very low density lipoprotein (VLDL) cholesterol after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Ratio | 0.92 (44.3) | 0.97 (42.1) | 0.91 (42.2)

24. Secondary Outcome: Triglycerides as a Ratio to Baseline at 52 Weeks
Description: Triglycerides after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Ratio | 0.91 (48.3) | 0.96 (44.2) | 0.91 (44.0)

25. Secondary Outcome: Free Fatty Acids as a Ratio to Baseline at 52 Weeks
Description: Free fatty acids after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Ratio | 0.74 (60.8) | 0.70 (59.3) | 0.93 (49.5)

26. Secondary Outcome: Fasting C-peptide as a Ratio to Baseline at 52 Weeks
Description: Fasting C-peptide after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 272
Ratio | 0.61 (75.6) | 0.42 (82.6) | 1.12 (29.9)

27. Secondary Outcome: Fasting Human Insulin as a Ratio to Baseline at 52 Weeks
Description: Fasting human insulin after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Ratio | 0.90 (89.0) | 0.61 (81.1) | 1.52 (66.6)

28. Secondary Outcome: Fasting Glucagon as a Ratio to Baseline at 52 Weeks
Description: Fasting glucagon after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 272
Ratio | 0.95 (27.9) | 0.94 (27.6) | 0.96 (25.7)

29. Secondary Outcome: Proinsulin as a Ratio to Baseline at 52 Weeks
Description: Proinsulin after 52 weeks of treatment was represented as ratio to baseline (week 0) values.
Time Frame: After 52 weeks of treatment
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 270 | 266 | 264
Ratio | 0.18 (231.5) | 0.17 (188.8) | 0.59 (85.9)

30. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: Treatment emergent adverse event is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product. If the event had onset date before the first day of exposure on randomised treatment and increased in severity during the treatment period and until 7 days after the last drug date, then this event was considered as a TEAE.
Time Frame: 0-52 weeks
Population: as for outcome 3
Measure: Number; unit: Events
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Events | 873 | 829 | 885

31. Secondary Outcome: Number of Treatment Emergent Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  Severe hypoglycaemia according to the ADA definition: an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: 0-52 weeks
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Episodes | 135 | 362 | 136

32. Secondary Outcome: Number of Treatment Emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product. Nocturnal period: The period between 00:01 and 05:59 a.m. (both inclusive).
  Severe or BG confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification or BG confirmed by a plasma glucose value < 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
  Severe hypoglycaemia according to the ADA definition: an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. Plasma glucose concentrations may not be available during an event, but neurological recovery following the return of plasma glucose to normal is considered sufficient evidence that the event was induced by a low plasma glucose concentration.
Time Frame: 0-52 weeks
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Episodes | 16 | 42 | 0

33. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to American Diabetes Association (ADA) Definition
Description: Results represent total number of treatment emergent hypoglycaemic episodes that fall under ADA's definition of hypoglycaemia. ADA's definition of hypoglycaemia includes following categories:
  1. Severe hypoglycaemia
  2. Documented symptomatic hypoglycaemia
  3. Asymptomatic hypoglycaemia
  4. Probable symptomatic hypoglycaemia
  5. Pseudo-hypoglycaemia. Treatment emergent hypoglycaemic episode is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
Time Frame: 0-52 weeks
Population: as for outcome 3
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Episodes | 4830 | 6340 | 162

34. Secondary Outcome: Anti-drug Antibodies: Anti-insulin Degludec Antibodies
Description: Insulin degludec (IDeg)-specific antibodies were measured at week 52, as %B/T (percentage of bound & precipitated radioactive drug/total added drug to the sample). A sample is measured in 2 different series. In series 1, the radioactive IDeg (tracer) and surplus unlabeled IDeg are added to the sample. In series 2, the tracer and surplus unlabeled human insulin are added to the sample. Series 1 represents unspecific background binding. Series 2 represents IDeg specific antibodies including unspecific background binding. The reported %B/T is calculated by subtracting the background %B/T in series 1 from the %B/T result in series 2. If the background result has higher values than the %B/T in series 2, the resulting value is negative %B/T. Here, a negative %B/T value means that the test samples do not have IDeg-specific antibodies. The reason for getting a negative value for %B/T is due to variation in the analytical background. Thus, the results presented are not a change from baseline.
Time Frame: at week 52
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (819 subjects). Subjects in the safety set contributed to the evaluation "as treated". Missing data were imputed using LOCF method. This endpoint is only applicable for subjects in IDegLira and IDeg arm.
Measure: Mean (Standard Deviation); unit: Percentage B/T
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 275 | 271
Percentage B/T | 0.12 (3.34) | -0.11 (0.42)

35. Secondary Outcome: Anti-drug Antibodies: Number of Participants Positive or Negative for Anti-liraglutide Antibodies
Description: Anti-liraglutide antibodies were measured at week 52. Number of participants positive or negative for anti-liraglutide antibodies at week 52 were reported.
Time Frame: at week 52
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (819 subjects). Subjects in the safety set contributed to the evaluation "as treated". Missing data were imputed using LOCF method.This endpoint is only applicable for subjects in IDegLira and Lira arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Liraglutide
Number analyzed (Participants) | 275 | 273
Participants
  Negative | 247 | 224
  Positive | 28 | 49

36. Secondary Outcome: Change in Clinical Evaluation: Fundoscopy or Fundus Photography
Description: The result of the fundus photography/dilated fundoscopy was interpreted by the investigator into following categories: Normal; Abnormal (Abn), Not Clinically significant (NCS); Abnormal, Clinically significant (CS). Reported results are number of subjects with 'normal'; 'Abn, NCS' and 'Abn, CS' fundoscopy/fundus photography results at screening (week -2 to week 0) and week 52.
Time Frame: at screening (week -2 to week 0), at week 52
Population: Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparator (819 subjects). Subjects in the safety set contributed to the evaluation "as treated". Number Analyzed = subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Participants
  Left eye - at screening visit - normal: number analyzed (Participants) | 274 | 271 | 272
  Left eye - at screening visit - normal | 225 | 213 | 211
  Left eye - at screening visit - Abn, NCS: number analyzed (Participants) | 274 | 271 | 272
  Left eye - at screening visit - Abn, NCS | 10 | 16 | 14
  Left eye - at screening visit - Abn, CS: number analyzed (Participants) | 274 | 271 | 272
  Left eye - at screening visit - Abn, CS | 39 | 42 | 47
  Left eye - week 52 - normal: number analyzed (Participants) | 274 | 271 | 272
  Left eye - week 52 - normal | 217 | 214 | 212
  Left eye - week 52 - Abn, NCS: number analyzed (Participants) | 274 | 271 | 272
  Left eye - week 52 - Abn, NCS | 17 | 16 | 15
  Left eye - week 52 - Abn, CS: number analyzed (Participants) | 274 | 271 | 272
  Left eye - week 52 - Abn, CS | 40 | 41 | 45
  Right eye - at screening visit - normal | 224 | 212 | 207
  Right eye - at screening visit - Abn, NCS | 10 | 14 | 12
  Right eye - at screening visit - Abn, CS | 41 | 45 | 54
  Right eye - week 52 - normal | 220 | 217 | 209
  Right eye - week 52 - Abn, NCS | 14 | 14 | 15
  Right eye - week 52 - Abn, CS | 41 | 40 | 49

37. Secondary Outcome: Change in Clinical Evaluation: Electrocardiogram (ECG)
Description: The result of the ECG was interpreted by the investigator into following categories: Normal; Abnormal (Abn), Not Clinically significant (NCS); Abnormal, Clinically significant (CS). Reported results are number of subjects with 'normal'; 'Abn, NCS' and 'Abn, CS' ECG results at screening (week -2 to week 0) and week 52.
Time Frame: at screening (week -2 to week 0), at week 52
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
Participants
  At screening visit - normal | 228 | 230 | 222
  At screening visit - Abn, NCS | 40 | 38 | 41
  At screening visit - Abn, CS | 7 | 3 | 10
  Week 52 - normal | 238 | 232 | 233
  Week 52 - Abn, NCS | 30 | 35 | 34
  Week 52 - Abn, CS | 7 | 4 | 6

38. Secondary Outcome: Change in Clinical Evaluation: Pulse
Description: Change in pulse after 52 weeks of treatment.
Time Frame: Week 0, week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
Number analyzed (Participants) | 275 | 271 | 273
beats per minute | 3.9 (9.5) | 0.8 (8.9) | 4.2 (9.1)

39. Secondary Outcome: Serum Concentrations of Insulin Degludec
Description: Samples from the IDegLira and IDeg arms were analysed for serum concentrations of insulin degludec using validated ELISA assays.
Time Frame: Weeks 2, 8, 16, 26, 44, 52
Population: Full Analysis Set (FAS) included all randomised subjects (819 subjects). All subjects in FAS with at least one valid concentration value were included in the analysis. No imputations of missing concentration values were applied. Number Analyzed = subjects with available data. This endpoint is only applicable for subjects in IDegLira and IDeg arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 275 | 271
pmol/L
  At week 2: number analyzed (Participants) | 274 | 270
  At week 2 | 1468.7 (55.9) | 1477.1 (61.3)
  At week 8: number analyzed (Participants) | 271 | 267
  At week 8 | 2246.0 (72.2) | 2524.6 (71.5)
  At week 16: number analyzed (Participants) | 264 | 262
  At week 16 | 2511.0 (83.6) | 2856.4 (84.4)
  At week 26: number analyzed (Participants) | 264 | 256
  At week 26 | 2597.3 (88.3) | 2946.9 (91.1)
  At week 44: number analyzed (Participants) | 254 | 248
  At week 44 | 2766.6 (85.8) | 3238.8 (91.7)
  At week 52: number analyzed (Participants) | 270 | 266
  At week 52 | 2393.8 (116.7) | 3124.4 (101.2)

40. Secondary Outcome: Plasma Concentrations of Liraglutide
Description: Samples from the IDegLira and liraglutide arms were assayed for plasma concentrations of liraglutide using validated ELISA assays.
Time Frame: Weeks 2, 8, 16, 26, 44, 52
Population: Full Analysis Set (FAS) included all randomised subjects (819 subjects). All subjects in FAS with at least one valid concentration value were included in the analysis. No imputations of missing concentration values were applied. Number Analyzed = subjects with available data. This endpoint is only applicable for subjects in IDegLira and Lira arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pmol/L
Arm/Group | Insulin Degludec/Liraglutide | Liraglutide
Number analyzed (Participants) | 275 | 273
pmol/L
  At week 2: number analyzed (Participants) | 274 | 270
  At week 2 | 5681.3 (49.4) | 6081.6 (65.4)
  At week 8: number analyzed (Participants) | 271 | 270
  At week 8 | 9107.8 (61.4) | 14539.5 (71.0)
  At week 16: number analyzed (Participants) | 262 | 268
  At week 16 | 10038.1 (69.5) | 14046.5 (73.0)
  At week 26: number analyzed (Participants) | 264 | 267
  At week 26 | 9995.3 (77.5) | 13904.2 (91.8)
  At week 44: number analyzed (Participants) | 253 | 262
  At week 44 | 8791.7 (81.0) | 12855.6 (112.7)
  At week 52: number analyzed (Participants) | 269 | 269
  At week 52 | 7426.2 (103.5) | 12127.4 (142.4)

ADVERSE EVENTS:
Time Frame: Week 0 (randomisation) to week 52 (end of treatment) and 7 days after end of treatment.
Description: Treatment emergent adverse event is defined as an event that had onset date on or after the first day of trial product administration, and no later than 7 days after the last day on trial product.
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Liraglutide
All-Cause Mortality (participants affected / at risk) | 1/275 | 0/271 | 0/273
Serious Adverse Events (participants affected / at risk) | 17/275 | 13/271 | 14/273
Other Adverse Events (participants affected / at risk) | 153/275 | 137/271 | 158/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=275) | Insulin Degludec (N=271) | Liraglutide (N=273)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Large intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thrombotic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=275) | Insulin Degludec (N=271) | Liraglutide (N=273)
Constipation (Gastrointestinal disorders) | 27 (28) | 12 (12) | 38 (42)
Diabetic retinopathy (Eye disorders) | 17 (17) | 12 (14) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 15 (20) | 12 (14) | 24 (31)
Eczema (Skin and subcutaneous tissue disorders) | 16 (18) | 6 (6) | 9 (10)
Headache (Nervous system disorders) | 7 (11) | 7 (12) | 15 (17)
Influenza (Infections and infestations) | 15 (15) | 9 (9) | 9 (9)
Lipase increased (Investigations) | 6 (8) | 0 (0) | 15 (15)
Nausea (Gastrointestinal disorders) | 9 (13) | 5 (7) | 23 (30)
Pharyngitis (Infections and infestations) | 11 (13) | 15 (18) | 9 (9)
Viral upper respiratory tract infection (Infections and infestations) | 106 (166) | 91 (161) | 94 (155)
Weight increased (Investigations) | 4 (4) | 19 (19) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT02607306/Prot_SAP_000.pdf